CLINICAL TRIAL: NCT03790423
Title: Phase I: PET Imaging of Tissue Factor (TF) Expression in Patients With Primary and Metastastic Cancer Using 18F-ASIS.
Brief Title: 18F-ASIS PET/CT Imaging of Tissue Factor Expression In Patients With Primary and Metastastic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mathias Dyrberg Loft, Principal Investigator, MD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AK2018_1; 2015-005583-42 (EudraCT Number)
Record Dates: First submitted 2018-12-20; First posted 2018-12-31 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer; Lung Cancer; Pancreatic Cancer; Ovarian Cancer; Cervix Cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-ASIS PET (Experimental): One injection of 18F-ASIS (app. 200 MBq) followed by 3 PET/CT scans 1 hour, 2 hours and 4hours post-injection
  Interventions: Drug: Injection of 18F-ASIS; Other: PET/CT scan

INTERVENTIONS:
Drug: Injection of 18F-ASIS — Each patient will receive one injection of 18F-ASIS (approximately 200 Mbq)
Other: PET/CT scan — Following one injection of 18F-ASIS the patients will be PET/CT scanned at 1 hour, 2 hours and 4 hours post-injection

SUMMARY:
The primary objective of the trial is to test the new radio tracer 18F-ASIS for PET imaging of tissue factor (TF) expression. The tracer has the potential of identifying tumors with high levels of TF expression, which is expected to correlate with tumor aggression and prognosis. Furthermore, the tracer can potentially be used as companion imaging diagnostic agent for identifying patients eligible for TF directed therapies.

This is a first-in-man study to test the radio tracer in cancer patients. Safety, biodistribution and dosimetry will be evaluated by repeated PET imaging (1 hour, 2 hours and 4 hours post-injection).

DETAILED DESCRIPTION:
The primary objective of the trial is to test the new radio tracer 18F-ASIS for PET imaging of tissue factor (TF) expression. The tracer has the potential of identifying tumors with high levels of TF expression, which is expected to correlate with tumor aggression and prognosis. Furthermore, the tracer can potentially be used as companion imaging diagnostic agent for identifying patients eligible for TF directed therapies.

This is a first-in-man study to test the radio tracer in cancer patients. Safety, biodistribution and dosimetry will be evaluated by repeated PET imaging (1 hour, 2 hours and 4 hours post-injection).

The primary end points are safety, biodistribution and dosimetry of 18F-ASIS. In addition, the quantitative uptake of 18F-ASIS will be compared to the expression of TF measured directly in tumor tissue obtained by surgery or biopsies. The study will be monitored and evaluated in accordance with the principles of Good Clinical Practice (GCP).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast, lung, pancreatic, cervix or ovarian cancer
* Capable of understanding the patient information in Danish and giving full informed consent

Exclusion Criteria:

* Pregnancy
* Breast-feeding
* Weight above 140 kg
* History of allergic reaction attributable to compounds of similar chemical or biologic composition to 18F-ASIS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
1.Biodistribution of the radiotracer 18F-ASIS estimated by PET | 4 hours
  The biodistribution of the 18F-ASIS radiotracer estimated from the standardized uptake values (SUV) of the major organs obtained from the patient's repeated PET imaging with the radiotracer 18F-ASIS
2.Dosimetry of the radiotracer 18F-ASIS estimated by PET | 4 hours
  Dosimetry will be calculated with the use of OLINDA/EXM software (mSv) based on repeated PET imaging with the radiotracer 18F-ASIS
3. Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 48 hours
  The safety of 18F-ASIS PET as measured by the number of participants with adverse events within 48 hours following the 18F-ASIS PET assessed by CTCAE v5.0

SECONDARY OUTCOMES:
1.Quantitative uptake of the radiotracer 18F-ASIS in tumor tissue | 4 hours
  The patients will be PET scanned 1 hour, 2 hours and 4 hours post-injection of the radiotracer 18F-ASIS. These timepoints will be used for assessment of tumor uptake by the use of maximum and mean standardized uptake value (SUV).

CONTACTS AND LOCATIONS:
Overall Officials: Mathias D Loft, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark